CLINICAL TRIAL: NCT03567031
Title: Impact of CO2 on Cerebral Blood Flow in Infants Less Than 6 Months During General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Bruno Greff, Principal Investigator, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #2017-1309
Record Dates: First submitted 2018-05-23; First posted 2018-06-25 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia, General; Infant
Keywords: Pediatric Anesthesia; Near-Infrared Spectroscopy; End-Tidal CO2; Cerebral Blood Flow

STUDY DESIGN:
Intervention Model Description: Cerebral blood flow is measured in each patient at 3 different, controlled levels of end-tidal CO2
Masking Description: Patient is under general anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Arm (Experimental): In each patient, under ongoing standard general anesthesia in a stable state, EtCO2 is manually modified to reach predefined values, and after waiting until cerebral blood flow has reached steady state, NIRS and DTC values are noted.
  Interventions: Procedure: EtCO2 modification

INTERVENTIONS:
Procedure: EtCO2 modification — Controlled modification of EtCO2 through modification of ventilation parameters under general anesthesia without spontaneous breathing

SUMMARY:
The study aims at assessing cerebral blood flow variations following expired CO2 variations in anaesthetized infants less than 6 months, during a routine general anesthesia.

DETAILED DESCRIPTION:
The study aims at assessing cerebral blood flow (measured with Near-Infrared Reflectance Spectroscopy - NIRS - and transcranial Doppler - DTC) variations following end-tidal expired CO2 variations in anaesthetized infants less than 6 months, during a routine general anesthesia performed according to standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Age < or = 6 months
* ASA class < or = 3
* General anesthesia required for surgery

Exclusion Criteria:

* No parental consent
* Emergency surgery
* Preexisting neurological condition
* Hemodynamic instability
* Preexisting hypoxemia and/or hypercapnia
* Laparoscopy or thoracoscopy, if expected EtCO2 level achieving would require unsafe ventilation parameters

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
NIRS variation | 5 to 10 minutes
  Near-Infrared Spectroscopy value variation after EtCO2 modification

SECONDARY OUTCOMES:
DTC variation | 5 to 10 minutes
  Transcranial Doppler values variation after EtCO2 modification

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Greff, MD, Principal Investigator — Sainte Justine's Hospital; Ossam Rhondali, MD, Study Director — Sainte Justine's Hospital; Jose Luis Martinez, MD, Study Chair — Sainte Justine's Hospital; Chantal Crochetière, MD, Study Chair — Sainte Justine's Hospital; Valérie Gaspard, MD, Study Chair — Sainte Justine's Hospital
Locations (1):
- Sainte Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT03567031/Prot_ICF_000.pdf